## **The Strategy of Prednisone Reduction**

For

TACTIC-SS - A Pilot Study in Severe Patients with Takayasu Arteritis.

Clinical Trial No.: NCT04300686

Department of Rheumatology

Zhongshan Hospital, Fudan University

Date: 2020-11-10

- 1. All the enrolled patients in TACTIC-SS were prescribed the strategy prednisone and methotrexate, as well as the biological agents adalimumab or tocilizumab according to the randomized group.
- 2. The dose of methotrexate is 15mg per week. The adalimumab is 40mg.q2weeks.IH, while the tocilizumab is 8mg/Kg. qm.IH.
- 3. The dose of prednisone was adjusted according to the following schedule.
- 4. The disease remission was defined as the disease status turning to inactivity.

## **Background glucocorticoid treatment (Routine Protocol)**

| | | Prior prednisone | Prior prednisone | Prior prednisone Notes |
|---|---|---|---|---|
| | | less than 40mg.qd | more than | less than 40mg.qd |
| | | (active status) | 40mg.qd | (inactive) or |
| | | , | | complicated with |
| | | | | infection |
| months | weeks | Dose | Dose | Dose |
| 0 | 0 | 40 | 40 | 30 |
| 1 | 2 | 35 | 35 | 30 |
| 1 | 4 | 30 | 30 | 25 |
| 2 | 6 | 25 | 25 | 25 |
| 2 | 8 | 20 | 20 | 25 |
| 3 | 12 | 15 | 15 | 20 |
| 4 | 16 | 10 | 10 | 15 |
| 5 | 20 | 10 | 10 | 10 |
| 6 | 24 | 10 | 10 | 10 |
| Biological agents switched if the disease remission was not achieved, and the prednisone would return | | | | |
| to 40mg. | | | | |
| 7 | 28 | 10 | 10 | 10 |
| 8 | 32 | 5 | 5 | 5 |
| 9 | 36 | 5 | 5 | 5 |
| 10 | 40 | 5 | 5 | 5 |
| 11 | 44 | 5 | 5 | 5 |
| 12 | 48 | 2.5 | 2.5 | 2.5 |
| Extended follow-up with prednisone free. If relapse occurred during follow-up, patients exited the | | | | |
| investigation. | | | | |
| 13 | 52 | 2.5 | 2.5 | 2.5 |
| 14 | 56 | 2.5 | 2.5 | 2.5 |
| 15 | 60 | 0 | 0 | 0 |
| 16 | 64 | 0 | 0 | 0 |
| 17 | 68 | 0 | 0 | 0 |
| 18 | 72 | | | |

## Notes:

Prednisone adjustment for special conditions.

- 1. If infection occurs (antibiotics needed), the prednisone would sustain the current dose and would not decrease till next month. Correspondingly, the biological agents would also suspend for a month as well.
- 2. After the initial 6 months' treatment, the biological agent strategy would be switched to the opposite if the disease remission could not be achieved, and the prednisone would return to 40mg as well.
- 3. The target dose of prednisone is 0 mg at the 48-week. Subsequently, patients would be followed up with prednisone free for another 6 months. If relapse occurred during this period, patients would exit the study immediately.